CLINICAL TRIAL: NCT00357708
Title: A Phase I Trial of SAHA (NSC 701852) and Decitabine (IND 50733, NSC 127716) in Patients With Relapsed, Refractory or Poor Prognosis Leukemia
Brief Title: Vorinostat and Decitabine in Treating Patients With Relapsed, Refractory, or Poor-Prognosis Hematologic Cancer or Other Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03088; 2005-0723; U01CA062461 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Chronic Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Philadelphia Chromosome Negative Chronic Myelogenous Leukemia; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Decitabine; Vorinostat

ARMS (1):
- Treatment (decitabine, vorinostat) (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 and oral vorinostat (SAHA) three times daily on days 6-19. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 6 patients receive escalating doses of decitabine and SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at that dose.
  Interventions: Drug: decitabine; Drug: vorinostat; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat and decitabine in treating patients with relapsed, refractory, or poor-prognosis hematologic cancer or other diseases. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with decitabine may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerated dose (MTD) and dose limiting toxicities (DLT) of vorinostat in combination with Decitabine in patients with relapsed/refractory or poor prognosis acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), myelodysplastic syndrome (MDS) or chronic myeloid leukemia in accelerated or blastic phase (CML-BP).

1.2 To describe the clinical activity of the combination of Decitabine and vorinostat in this patient population.

1.3 To determine the in vivo molecular effects of this combination. This will include measuring the effects on DNA methylation, histone H3 and H4 acetylation and changes in gene expression.

1.4 To determine the pharmacokinetic characteristics of the combination.

OUTLINE: This is a dose-escalation study.

Patients receive decitabine IV over 1 hour on days 1-5 and oral vorinostat (SAHA) three times daily on days 6-19. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of decitabine and SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at that dose.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), chronic myelogenous leukemia (CML), myelodysplastic syndrome (MDS) or myeloproliferative disease (MPD)
* Patients with refractory or relapsed acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), chronic myelogenous leukemia (CML), myelodysplastic syndrome (MDS) IPSS intermediate 1 and above and myeloproliferative disease (MPD) will be considered for the study; patients with CML are eligible if they have documented hematologic resistance to imatinib mesylate, or lack of any cytogenetic response to imatinib mesylate after 12 months of therapy; patients with Chronic Myelomonocytic Leukemia (CMML) or Philadelphia negative CML are eligible if their disease is not controlled by standard therapy (e.g. hydroxyurea) or if they show signs of disease progression on standard therapy (blast count > 5%, platelet count < 100K); patients with Acute Promyelocytic Leukemia are eligible only if they have progressed after standard chemotherapy, ATRA as well as Arsenic Trioxide therapy; untreated patients older than 60 years of age with AML (except APL) or MDS IPSS intermediate 1 and above, not eligible for standard therapy, are also eligible
* Patients must have been off chemotherapy for 2 weeks (six weeks for nitrosoureas or mitomycin C) prior to entering this study and recovered from the toxic effects of that therapy unless there is evidence of rapidly progressive disease; if there is evidence or rapidly progressive disease, the use of hydroxyurea is allowed prior to starting the clinical trial and during the first cycle of therapy; other histone deacetylase inhibitors, including valproic acid, should be stopped 2 weeks prior to entering this study
* Life expectancy of greater than 8 weeks
* ECOG performance status 0-2
* Total bilirubin =< 2 mg/dL
* AST(SGOT) or ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine =< 2 mg/dL
* Cardiac ejection fraction >= 50%
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with clinical evidence of CNS disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or decitabine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat
* HIV-positive patients receiving combination antiretroviral therapy are ineligible
* Vorinostat should not be taken concomitantly with other HDAC inhibitors or compounds with HDAC inhibitor like activity, such as valproic acid; patients who have received such agents as anti-tumor therapy should not enroll in vorinostat oncology trials; patients who have received such agents for other indications, e.g. epilepsy, may enroll on vorinostat trials after a 30 day washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of vorinostat and decitabine | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Issa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bernot KM, Siebenaler RF, Whitman SP, Zorko NA, Marcucci GG, Santhanam R, Ahmed EH, Ngangana M, McConnell KK, Nemer JS, Brook DL, Kulp SK, Chen CS, Frankhouser D, Yan P, Bundschuh R, Zhang X, Dorrance AM, Dickerson KE, Jarjoura D, Blum W, Marcucci G, Caligiuri MA. Toward personalized therapy in AML: in vivo benefit of targeting aberrant epigenetics in MLL-PTD-associated AML. Leukemia. 2013 Dec;27(12):2379-82. doi: 10.1038/leu.2013.147. Epub 2013 May 10. No abstract available. PMID 23660685